CLINICAL TRIAL: NCT06387888
Title: The Effect of Mother's Voice on the Levels of Pain and Comfort in Newborns on Mechanical Ventilation: a Randomized Controlled Study
Brief Title: The Effect of Mother's Voice on the Levels of Pain and Comfort in Newborns
Acronym: Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aysel kokcudogan, Assistant professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-31034136-302.08.01-4221
Record Dates: First submitted 2024-04-20; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Newborns
Keywords: Comfort,; Mechanical ventilatör,; Mother's voice,; Newborn,; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group-30 (Experimental): During the care, from the beginning to the end, mother's voice was played to the newborns. It took about 20 minutes. The mini Bluetooth speaker and the decibel meter were disinfected with the rapid surface disinfectant used in the clinic. The speaker was placed 30 cm away from the infant's ear and the sound level in the incubator was adjusted to be 50-60 dB by using a decibel meter. Mother's voice was played from the beginning of the provision of care and continued for 15 minutes after the end of the provision of care. During the provision of care, COMFORTneo scores, pain scores, and vital signs were measured and recorded on the vital signs follow-up form.
  Interventions: Other: Listening to mother's voice
- Control group-30 (No Intervention): Standard nursing care lasting 20 minutes was performed in the routine sound environment of the neonatal intensive care unit. COMFORTneo scores, pain scores, and vital signs were measured and recorded on the vital signs follow-up form.

INTERVENTIONS:
Other: Listening to mother's voice — During the care, from the beginning to the end, mother's voice was played to the newborns. It took about 20 minutes. The mini Bluetooth speaker and the decibel meter were disinfected with the rapid surface disinfectant used in the clinic. The speaker was placed 30 cm away from the infant's ear and the sound level in the incubator was adjusted to be 50-60 dB by using a decibel meter (Official Gazette, 2018). Mother's voice was played from the beginning of the provision of care and continued for 15 minutes after the end of the provision of care. During the provision of care, COMFORTneo scores, pain scores, and vital signs were measured and recorded on the vital signs follow-up form.
  Arms: Intervention group-30

SUMMARY:
This study was conducted in a randomized controlled experimental type to determine the effect of maternal voice during care on pain and comfort level in term newborns receiving mechanical ventilation. The sample of the study was consisted of 60 term newborns receiving mechanical ventilation who were hospitalized in the 7-bed Neonatal Intensive Care Unit of a private hospital in Istanbul in accordance with the selection criteria. Introductory Information Form, Vital Signs Follow-up Form, Neonatal Comfort Behavior Scale and Neonatal Pain Scale (NPASS) forms prepared by the researchers were used as data collection tools.

DETAILED DESCRIPTION:
Intervention group: During the care, from the beginning to the end, mother's voice was played to the newborns. It took about 20 minutes. The mini Bluetooth speaker and the decibel meter were disinfected with the rapid surface disinfectant used in the clinic. The speaker was placed 30 cm away from the infant's ear and the sound level in the incubator was adjusted to be 50-60 dB by using a decibel meter Mother's voice was played from the beginning of the provision of care and continued for 15 minutes after the end of the provision of care. During the provision of care, COMFORTneo scores, pain scores, and vital signs were measured and recorded on the vital signs follow-up form.

Control group: Standard nursing care lasting 20 minutes was performed in the routine sound environment of the neonatal intensive care unit. COMFORTneo scores, pain scores, and vital signs were measured and recorded on the vital signs follow-up form.

ELIGIBILITY:
Inclusion Criteria:

* Connected to a mechanical ventilator (intubation or nasal CPAP),
* Term newborns (born at 37-42 weeks),
* No neurological disorders,
* No congenital or acquired hearing malformations,
* The family consents for their infant to participate in the study,

Exclusion Criteria:

* Diagnosis of asphyxia,
* Use of sedatives or analgesics,
* Congenital anomaly,
* Underwent an extra invasive procedure or surgical intervention,
* Parents with congenital hearing problems.

Ages: 3 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Comfort Behavior Scale | 20 minutes
  The scale is for 0-100-day-old infants and term or preterm newborns experiencing acute or chronic pain and treated with or without mechanical ventilation.

SECONDARY OUTCOMES:
Neonatal Comfort Behavior Scale (COMFORTneo): | 20 minutes
  COMFORTneo consists of 7 items on alertness, calmness/agitation, respiratory response, crying, body movement, facial tension, and muscle tone. Of these items, "respiratory response" is evaluated in newborns on mechanical ventilation and "crying" is evaluated in spontaneously breathing newborns.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Kökcü Doğan, Study Director — Istanbul Medipol University Hospital
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Beykoz, Turkey (Türkiye)